CLINICAL TRIAL: NCT01676883
Title: Plantar Callosities and the Validity of Body Composition Assessment by Bio-impedance in Severely Obese Persons
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2012/1018
Record Dates: First submitted 2012-08-29; First posted 2012-08-31 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2016-06

CONDITIONS: Obesity, Morbid
Keywords: Body constitution; Anthropometry; Electric impedance
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- body composition assessment (Experimental): Bioelectric impedance measurement pre- and post removal of calluses and corns (pedicure), then air-displacement plethysmography (gold standard)
  Interventions: Device: Bioelectric impedance; Device: Air displacement plethysmography

INTERVENTIONS:
Device: Bioelectric impedance — removal of calluses and corns by pedicure
  Other Names: BIA
Device: Air displacement plethysmography
  Other Names: ADP

SUMMARY:
Studies have confirmed the association between plantar callosities and severely obese individuals. Bioelectrical impedance analysis (BIA) is an increasingly popular tool for estimating body composition because it is easy to use, noninvasive, relatively inexpensive, and can be performed across a wide range of subjects.

Our hypotheses for this study are: (1)plantar callosities influence the body composition measurements obtained by bioelectrical impedance analysis BIA, and (2) BIA underestimates the percentage of body fat compared with air-displacement plethysmography (BodPod).

DETAILED DESCRIPTION:
As the prevalence of obesity continues to increase, many parts of the world are progressively facing a rise in the number of people who fall under WHO obesity class 2 and 3. Since severe obesity is characterized by large alterations in body compartments when compared to overweight or non-obese individuals, there is a need for the evaluation of the body composition of severely obese persons. There is very few published research available on what methods of body composition measurements can be used on this population.

Other studies have also shown the tendency of bioelectrical impedance analysis (BIA) instruments to underestimate percentage of fat mass and overestimate the percentage of fat free nass, compared with gold-standard techniques. We think that plantar callosities might have contributed to the lack of accurate measurements. Thus, the primary aim of this study is to determine whether plantar callosities influence the validity of body composition measurements obtained by BIA, using the InBody 720. The secondary aim is to assess the validity of the body composition measurements obtained by BIA (InBody 720) in severely obese individuals, using air-displacement plethysmography (BodPod) as the gold standard. Additionally, we will explore various sources of error using test-retest reliabilities by measuring body composition with different arm postures. We will examine this further to rule out the possibility of "positions of measurement" as a potential confounder of this study.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18-50 years old)
* class 2 and 3 obesity (BMI > 35 kg/m2)
* moderate to severe callosities

Exclusion Criteria:

* Intractable plantar keratosis (IPK), which are painful plantar calluses located under the metatarsal heads.
* pregnancy
* menopause
* diseases that cause water retention (edema, renal insufficiency, hypertension, etc.)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2012-10; Primary Completion 2013-03 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Body composition | 1 day
  Bioelectric impedance (using InBody 720) at three standardized arm postures angled at 15, 45 and 90 degrees, in randomized order; Air displacement plethysmography (ADP,using BodPod)

CONTACTS AND LOCATIONS:
Overall Officials: Bård Kulseng, MD PhD, Study Director — St. Olavs Hospital
Locations (1):
- Obesity policlinic of St. Olavs Hospital, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Roekenes J, Strommen M, Kulseng B, Martins C. The Impact of Feet Callosities, Arm Posture, and Usage of Electrolyte Wipes on Body Composition by Bioelectrical Impedance Analysis in Morbidly Obese Adults. Obes Facts. 2015;8(6):364-72. doi: 10.1159/000442033. Epub 2015 Nov 20. PMID 26584161